CLINICAL TRIAL: NCT04503616
Title: A Phase IB-II Study Of High-Dose Post-Transplant Cyclophosphamide, Abatacept, and Short-Duration Tacrolimus for the Prevention of Graft-Versus-Host Disease (GvHD) Following Haploidentical Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Cyclophosphamide, Abatacept, and Tacrolimus for GvHD Prevention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-00136
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Graft-versus-host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide; Abatacept; Tacrolimus

STUDY DESIGN:
Intervention Model Description: Interventional, non-randomized open label, 2- stage optimal Simon design with interim futility analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HSCT Patients (Experimental): Adult patients with hematological malignancies undergoing HLA-haploidentical HSCT from first-or second-degree family donors.
  Interventions: Drug: Cyclophosphamide, Abatacept, and Tacrolimus for GvHD Prevention

INTERVENTIONS:
Drug: Cyclophosphamide, Abatacept, and Tacrolimus for GvHD Prevention — Cyclophosphamide 50 mg/kg IV over 2 hours on Day +3 and +4 Abatacept 10 mg/kg IV on days +5, +14, and +28 Tacrolimus 0.02 mg/kg IV by continuous infusion, starting on day +5. May switch to oral when tolerated, adjusted to maintain a drug level between 5-12ng/mL. Treatment is discontinued on day +60 after a 4 week-taper

SUMMARY:
This is a single arm, open label, optimal 2-stage Simon design phase Ib-II clinical trial. Adult patients with hematological malignancies undergoing allogeneic HSCT from first- or second-degree haploidentical donor are eligible for the study if they meet the standard criteria defined in our institutional standard operation procedures (SOPs), meet all inclusion criteria, and do not satisfy any exclusion criteria. Patients will receive non-myeloablative, reduced-intensity or myeloablative conditioning regimen followed by peripheral blood hematopoietic stem cells. Patients will receive cyclophosphamide, abatacept, and short-duration tacrolimus for GvHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Karnofsky score ≥ 70%
3. No evidence of progressive bacterial, viral, or fungal infection
4. Creatinine clearance > 50 mL/min/1.72m2
5. Total bilirubin, ALT and AST < 2 x the upper limit of normal (except for diagnosed Gilbert's syndrome)
6. Alkaline phosphatase ≤ 250 IU/L
7. Left Ventricular Ejection Fraction (LVEF) > 45%
8. Adjusted Carbon Monoxide Diffusing Capacity (DLCO) > 60%
9. Negative HIV serology
10. Negative pregnancy test: confirmation per negative serum β-human chorionic gonadotropin (β-hCG) for women of childbearing age and potential.

Exclusion Criteria:

1. Donors are excluded in case of donor-specific HLA antibodies or positive cross-match.
2. Pregnant or nursing females or women of child bearing age or potential, who are unwilling to completely abstain from heterosexual sex or practice 2 effective methods of contraception from the first dose of conditioning regimen through day +180. A woman of reproductive capability is one who has not undergone a hysterectomy (removal of the womb), has not had both ovaries removed, or has not been post-menopausal (stopped menstrual periods) for more than 24 months in a row.
3. Male subjects who refuse to practice effective barrier contraception during the entire study treatment period and through a minimum of 90 days after the last dose of study drug, or completely abstain from heterosexual intercourse. This must be done even if they are surgically sterilized (i.e., post-vasectomy).
4. Inability to provide informed consent.
5. Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see Appendix E), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
6. Known allergies to any of the components of the investigational treatment regimen.
7. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
8. Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
9. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maher Abdul Hay, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Maher.Abdulhay@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Maher.Abdulhay@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Al-Homsi AS, Cirrone F, Wo S, Cole K, Suarez-Londono JA, Gardner SL, Hsu J, Stocker K, Bruno B, Goldberg JD, Levinson BA, Abdul-Hay M. PTCy, abatacept, and a short course of tacrolimus for GVHD prevention after haploidentical transplantation. Blood Adv. 2023 Jul 25;7(14):3604-3611. doi: 10.1182/bloodadvances.2023010545. PMID 37163349

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HSCT Patients
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HSCT Patients
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 60 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade II-IV Acute GvHD by Day +120
Description: The first day of grade II-IV acute GvHD will be used to calculate the cumulative incidence. The cumulative incidence will be defined as the percentage of participants with grade II-IV acute GvHD. The diagnosis of acute GvHD is based on clinical and pathological evaluation by the principal investigator in collaboration with the treating physician.
  Overall Grades of Acute GvHD:
  0 = none;
  1. = mild;
  2. = moderate;
  3. = severe;
  4. = life threatening
Time Frame: 120 days
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HSCT Patients
Number analyzed (Participants) | 46
Percentage of participants | 17.4 [9.2 to 32.9]

2. Secondary Outcome: Cumulative Incidence of Chronic GvHD
Description: The first day of chronic GvHD will be used to calculate the cumulative incidence of chronic GvHD. This endpoint will be evaluated through day +365 post-transplant.
Time Frame: Day 365
Reporting Status: Not Posted

3. Secondary Outcome: Cumulative Incidence of Primary Graft Failure
Description: Graft failure is defined as failure to achieve neutrophil engraftment by day +28 or lack of donor chimerism > 50% by day 45, not due to the underlying malignancy.
Time Frame: Day 45
Reporting Status: Not Posted

4. Secondary Outcome: Cumulative Incidence of Poor Graft Function
Description: Poor Graft Function defined by at least 2 of the following 3 criteria: Hemoglobin < 8 g/dL, ANC < 0.5 x 109/L, and platelets < 20 x 109/L. The cytopenia must be unexplained (such as by disease relapse) and unresponsive to cytokines and must last at least 4 weeks.
Time Frame: Day 28
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of Secondary Graft Failure
Description: Evaluated following engraftment through day +730. Secondary Graft Failure defined as poor graft function associated with donor chimerism < 5%.
Time Frame: Day 730
Reporting Status: Not Posted

6. Secondary Outcome: Number of Treatment-Related Deaths
Description: Number of participant deaths not attributable to disease relapse or progression. Will be evaluated to day +730.
Time Frame: Day 730
Reporting Status: Not Posted

7. Secondary Outcome: Relapse Rate
Description: Evaluated to day +730 and defined as the percentage of patients in whom the disease for which transplant is performed becomes evident by methods of disease detection after the transplant.
Time Frame: Day 730
Reporting Status: Not Posted

8. Secondary Outcome: GvHD and Relapse-Free Survival (GRFS)
Description: Evaluated to day +730 and defined as the percentage of participants who are without reported grade III-IV acute GvHD, without chronic GvHD requiring systemic therapy, and have not experienced relapse or death.
Time Frame: Day 730
Reporting Status: Not Posted

9. Secondary Outcome: Overall Survival
Description: Evaluated to day +730 and defined as percentage of participants alive at the end of the study's evaluation period.
Time Frame: Day 730
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 120 Days
Description: Collected during study visits and interviews of a study participant presenting for medical care, or upon review by a study monitor.
Arm/Group | HSCT Patients
All-Cause Mortality (participants affected / at risk) | 7/46
Serious Adverse Events (participants affected / at risk) | 19/46
Other Adverse Events (participants affected / at risk) | 24/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HSCT Patients (N=46)
Acute kidney injury (Renal and urinary disorders) | 5
Bacteremia (Infections and infestations) | 1
Blood bilirubin increased (Hepatobiliary disorders) | 3
Cytomegalovirus (CMV) reactivation (Infections and infestations) | 3
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Epstein-Barr Virus (EBV) reactivation (Infections and infestations) | 1
Febrile neutropenia (General disorders) | 6
Graft-versus-host disease (GvHD) (General disorders) | 1
Hematochezia with colostomy (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Meningitis (Infections and infestations) | 1
Multiorgan failture (General disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericardial tamponade (Cardiac disorders) | 1
Pulmonary airspace opacities (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Toxoplasmosis infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HSCT Patients (N=46)
Abdominal pain (Gastrointestinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 2
Bacteremia (Infections and infestations) | 4
Blood bilirubin increased (Hepatobiliary disorders) | 3
CMV reactivation (Infections and infestations) | 7
Colitis (Gastrointestinal disorders) | 1
Confusion (Nervous system disorders) | 1
Conjunctival hemorrhage (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increase (Renal and urinary disorders) | 1
Cytokine release syndrome (General disorders) | 1
Delirium (Nervous system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Dysuria (Renal and urinary disorders) | 2
EBV reactivation (Infections and infestations) | 1
Epitaxis (Blood and lymphatic system disorders) | 2
Facial nerve disorder (Nervous system disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 4
Flu like symptoms (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Hematuria (Renal and urinary disorders) | 2
Hypertension (Vascular disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Lethargy (Nervous system disorders) | 1
Mucositis (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 1
Papulopustular rash (Skin and subcutaneous tissue disorders) | 2
Pneumonia (Infections and infestations) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
Tremor (Nervous system disorders) | 1
Viremia (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT04503616/Prot_SAP_000.pdf